CLINICAL TRIAL: NCT05881239
Title: Digital Accessible Remote Olfactory Mediated Health Assessments for Preclinical AD
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Mark W Albers, Frank Wilkens and Family Endowed Scholar/ Asst. Prof. Neurology, Massachusetts General Hospital
Other Study IDs: 2022P002451
Record Dates: First submitted 2023-05-19; First posted 2023-05-31 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Subjective Cognitive Concerns; Mild Cognitive Impairment; Mild Behavioral Impairment; Healthy Aging
Keywords: Alzheimer's disease; Olfactory; Neurodegeneration; Mild Cognitive Impairment; Mild Behavioral Impairment; Subjective Cognitive Concerns; Olfactory dysfunction; Biomarker; Cognitive Assessment
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Anosmia; Nerve Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Subjective Cognitive Concerns (SCC): The composition of the proposed study population will reflect that of subjects recruited through the Longitudinal Cohort of the Massachusetts Alzheimer's Disease Research Center and that of patients treated by neurologists at the Memory and Movement Disorders Clinics at MGH as well as participants from the community.
  Interventions: Device: AROMHA Brain Health Test
- Mild Cognitive Impairment (MCI): The composition of the proposed study population will reflect that of subjects recruited through the Longitudinal Cohort of the Massachusetts Alzheimer's Disease Research Center and that of patients treated by neurologists at the Memory and Movement Disorders Clinics at MGH as well as participants from the community.
  Interventions: Device: AROMHA Brain Health Test
- Mild Behavioral Impairment [prominent apathy] (MBI): The composition of the proposed study population will reflect that of subjects recruited through the Longitudinal Cohort of the Massachusetts Alzheimer's Disease Research Center and that of patients treated by neurologists at the Memory and Movement Disorders Clinics at MGH as well as participants from the community.
  Interventions: Device: AROMHA Brain Health Test
- Age-matched Controls: We will utilize community sampling to recruit 100 age-matched controls.
  Interventions: Device: AROMHA Brain Health Test

INTERVENTIONS:
Device: AROMHA Brain Health Test — The AROMHA Brain Health Test is a self-administered, at-home smell test developed as a potential primary screen for identifying individuals at risk for developing Alzheimer's and as a means to follow disease progression in individuals without overt cognitive symptoms. The smell test device consists of five physical smell cards and a paired web-based app that directs participants on how to sample odors and asks them questions regarding what they have smelled. The 45-minute smell test battery includes measures of odor intensity, identification, memory, and discrimination.

SUMMARY:
The goal of this study is to objectively test one's sense of smell, called olfaction, in participants with Subjective Cognitive Concerns (SCC), Mild Cognitive Impairment, Mild Behavioral Impairment (MBI), and age-matched controls. The main question it aims to answer is whether the AROMHA Brain Health Test could serve as a predictive biomarker of neurodegenerative disorders. This understanding will aid in the development of a noninvasive, cost-effective diagnostic tool that reliably and specifically distinguishes disease and normal aging populations.

Participants will take the approximately 45-minute AROMHA Brain Health Smell Test where they will peel and sniff labels on the physical smell cards and answer questions on the web-based app relating to what they smelled. Participants will undergo tests for odor intensity, odor identification, odor discrimination, and episodic olfactory memory, but will not be provided the results of these tests.

ELIGIBILITY:
Inclusion Criteria:

* A clinical or research consensus diagnosis of the patient's condition or control status.
* Individuals that are at least 18 years of age at the time of enrollment.
* Individuals that are no older than 100 years of age at the time of enrollment.

Exclusion Criteria:

* Primary pulmonary disease such as severe emphysema or asthma not under good medical control.
* Current sinusitis, common cold, upper respiratory infection, or nasal polyps.
* Current or recent (past 6 months) alcohol or substance dependence. A prior history of alcohol or substance abuse will not be grounds for exclusion.
* Pregnancy.
* Severe cognitive dysfunction that would preclude completion of the olfactory testing.
* An adverse reaction to fragrances (ie. they trigger a severe asthmatic attack or nausea).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Subjective Cognitive Concerns (SCC),
  2. Mild Cognitive Impairment,
  3. Mild Behavioral Impairment,
  4. Healthy Age-matched Controls.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
AROMHA Brain Health Test | 1 hour
  The AROMHA Brain Health Test is a battery of 18 odors across 5 smell cards. The subject smells each odor label and is tested on odor intensity, identification, memory, and discrimination. An increased number of correct responses indicates a better sense of smell. We will evaluate MCI patients' performance against age-matched controls.

SECONDARY OUTCOMES:
AROMHA Brain Health Test | 1 hour
  The AROMHA Brain Health Test is a battery of 18 odors across 5 smell cards. The subject smells each odor label and is tested on odor intensity, identification, memory, and discrimination. An increased number of correct responses indicates a better sense of smell. We will evaluate MBI patients' performance against age-matched controls.

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Albers, MD PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States